CLINICAL TRIAL: NCT00304980
Title: Comparative Evaluation of the Safety and the Efficacy of Artemether + Lumefantrine (Coartem™) vs. Sulfadoxine + Pyrimethamine (SP) in Both HIV+ and HIV- Adults With Uncomplicated P. Falciparum Malaria in Zambia
Brief Title: Comparative Evaluation of the Safety and the Efficacy of 2 Antimalarials Depending on HIV Status
Status: Terminated | Phase: Not Applicable | Type: Interventional
Sponsor: Institute of Tropical Medicine, Belgium (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 02 52 5 406
Record Dates: First submitted 2006-03-20; First posted 2006-03-21 (Estimated); Last update posted 2010-09-14 (Estimated); Status verified 2010-09

CONDITIONS: Plasmodium Falciparum Malaria
MeSH Terms: conditions — Malaria, Falciparum | interventions — Artemether; Pyrimethamine

INTERVENTIONS:
Drug: ARTEMETHER + LUMEFANTRINE VS. SULFADOXINE + PYRIMETHAMINE

SUMMARY:
The purpose of this study is to determine the safety and efficacy of sulfadoxine-pyrimethamine (SP) versus artemether-lumefantrine (Coartem) when administered to HIV+ and HIV- patients with uncomplicated P. falciparum malaria. Patients will be randomised to one of the 2 treatment and followed up (until day 14 actively) for 45 days.

ELIGIBILITY:
Inclusion Criteria:

* Man and non-pregnant women aged between 15 and 50.
* P.falciparum mono-infection of at least 1,000 parasites/µl.
* Body temperature ≥ 37.5°C at the moment of enrolment or history of fever in the preceding 48 hrs.
* Consent from patient obtained.

Exclusion Criteria:

* Pregnancy.
* Severe P. falciparum malaria .
* Documented intake of SP or Coartem two weeks or less prior recruitment.
* Other cause(s) of fever.
* Evidence of underlying chronic diseases (cardiac, renal, hepatic, malnutrition).
* History of allergy to study drug, or known allergy to other Sulphur drugs such as co-trimoxazol.

Ages: 15 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 3000
Dates: Start 2003-03; Study Completion 2005-04

PRIMARY OUTCOMES:
PCR corrected clinical and parasitological outcome at day 45

SECONDARY OUTCOMES:
Tolerability
Clinical recovery

CONTACTS AND LOCATIONS:
Overall Officials: Umberto D'Alessandro, MD,MSc, PHD, Principal Investigator — Institute of Tropical Medicine Antwerp
Locations (1):
- Tropical Disease Research Center, Ndola, Cupperbelt, Zambia

REFERENCES:
- [Result] Van Geertruyden JP, Mulenga M, Mwananyanda L, Chalwe V, Moerman F, Chilengi R, Kasongo W, Van Overmeir C, Dujardin JC, Colebunders R, Kestens L, D'Alessandro U. HIV-1 immune suppression and antimalarial treatment outcome in Zambian adults with uncomplicated malaria. J Infect Dis. 2006 Oct 1;194(7):917-25. doi: 10.1086/507310. Epub 2006 Aug 29. PMID 16960779